CLINICAL TRIAL: NCT06168500
Title: Narrow Diameter Implants Versus Standard Diameter Implants With Simultaneous Bone Regeneration For The Treatment Of Atrophic Posterior Area
Brief Title: Narrow Implants Vs Standard Implants With Simultaneous GBR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Klockner Implant System S.A. (Unknown); Botiss Medical AG (Other)
Responsible Party: Principal Investigator, Rodrigo González Terrats, Doctor Dental Surgery, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER-ECL-2018-06
Record Dates: First submitted 2023-11-15; First posted 2023-12-13 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Narrow Implant; Dental Implant; Bone Regeneration
Keywords: Narrow Implant
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental)
  Interventions: Procedure: Test group; Procedure: Control group
- Control group (Experimental)
  Interventions: Procedure: Test group; Procedure: Control group

INTERVENTIONS:
Procedure: Test group — 3.0mm diameter implant
Procedure: Control group — 4.0 diameter implant + guided bone regeneration

SUMMARY:
NDI represent an advisable treatment option when the mesio-distal space is compromised. In a recent retrospective study with a follow-up of 8 years in which they wanted to evaluate the long-term survival, complications, peri-implant conditions, marginal bone loss, and patient satisfaction of fixed dental prostheses supported by NDI in the posterior area. They observe a survival rate of 97% and absence of prosthetic complications after the study period time. More recently, Souza et al. performed a prospective randomized split mouth study with 3 years follow-up with the aim of comparing marginal bone level, implant survival and success rates and prosthesis success rates of NDI and SDI placed in the posterior area of the mandible to support single prosthesis. They observed an implant survival rate of 100% for both groups at 1 and 3 years. The prosthesis success rate at 1 and 3 years was of 95.4% and 100%, respectively.

NDI present a high survival rate on the evaluated studies. Therefore, the aim of the first study is to compare the patient related outcomes, implants and prostheses success and survival rates of pure titanium NDI versus SDI with simultaneous bone regeneration in narrow alveolar ridges at posterior areas of the maxilla and the mandible.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* 18 years old
* Healthy periodontal status (absence of generalized probing pocket depth (PPD) <4mm)
* Oral hygiene levels (FMPS <20 and FMBS <20)

Site:

* Ridge width of >5mm and <6.5mm and minimum bone height of 10mm prior evaluation on a CBCT scan
* Presence of antagonistic natural tooth or fixed prosthetic restoration
* Presence of adjacent teeth
* One maxillary or mandibular premolars
* Minimum of 3mm of keratinized tissue over the bone crest (20)
* Bone regeneration within the limits of the prosthetic restoration.

Implants:

* Unitary prosthesis
* Screwed retained restorations

Exclusion Criteria:

Patients

* Presence of active chronic or aggressive periodontal disease
* Presence of systemic disease which contraindicate surgery (patients with an ASA ≥ 3)
* Drugs or medications which may alter the results (chronic intake of analgesic medication)
* Smokers (>10cig/day)
* Pregnant women
* History of head and neck radiotherapy.

Site

* Anterior area (from 1.3 to 2.3 and from 3.3 to 4.3) and molar area
* Previous guided bone regeneration
* Location where there is not sufficient restorative space (mesio-distally <8mm for every restoration unit and <5mm from the bone crest to the antagonist)
* Implant dehiscence of more than 2/3 of the implant.

Implant

* Implants which cannot be restored with a screwed restoration
* Implants which doesn't reach a manual implant stability
* implants which after placement doesn't reach a favourable position according to the restoration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Marginal bone level difference | The changes in MBL will be registered at 8 weeks, 6 months, 12 months, and 3 years.
  To assess the MBL, each radiograph must register the most coronal aspect of the bone crest (BC) at mesial and distal to the implant, the position of the implant shoulder (IS) and the first bone to implant contact (FBiC). The marginal bone crest level (MBL) will be measured by calculating the distance between BC and IS. MBL will be considered negative when position of BC is coronal to IS, positive when position BC is apical to IS.

SECONDARY OUTCOMES:
Patient related outcomes | At 1, 2 and 12 weeks
  - Level of discomfort - at 1-, 2- and 12-weeks post-surgery (VAS scale): 0 - 4 (being 0 no discomfort and 4 very severe discomfort)
Patient Related Outcomes | At 1, 2 and 12 weeks
  Willingness of undergoing same surgical procedure - at 1-, 2- and 12-weeks post-surgery (VAS scale): 0 - 4 (being 0 will never undergo this surgery again and 4 no problem to repeat this surgery)
Patient Related Outcomes | At 7 days
  - Level of pain perceived - during first 7 days after surgery (VAS scale): 0-100 (being 0 no pain and 100 intolerable pain)
Patient Related Outcomes | At 7 days
  Medication required: Number of ibuprofen tablets taken between the 2nd and the 7th day.
Implant survival criteria: | 12 months
  Defined as the implant being still in function
Implant success criteria: | 12 months
  Defined as absence of:
  * Persistent pain, foreign body sensation, and/or dysesthesia
  * Recurrent peri-implant infection with suppuration
  * Implant mobility
  * Continuous radiolucency around the implant
  * Clinical probing depth (CPD) ≥5 mm associated with bleeding/suppuration on probing (BoP/SoP).
Prosthesis success criteria | 12 months
  * Absence of prosthesis (crown or abutment) mobility
  * Number of maintenance visits
  * Crown screw loosening
  * Abutment screw loosening
  * Implant fracture
  * Crown screw fracture
  * Abutment screw fracture
  * Crown chipping.
Resonance frequency analysis | Implant surgery and after 12 months
  Resonance frequency analysis using Penguin ® will be measured immediately after implant placement, when taking implant impressions
Level of keratinized tissue surrounding the implants | 12 months
  Level of keratinized tissue will be measured from the gingival margin of the restored implant to the mucogingival line using a periodontal millimetre probe.
Peri-implant mucosal thickness using a millimetre probe | 12 months
Presence of post-surgical complications | At 1, 2 and 12 weeks
  Defined as absence of:
  * Infection/suppuration
  * Wound dehiscence
  * Implant failure
  * Post-op oedema
Presence of peri-implant health | At 12 weeks, 6 and 12 months
  Defined as:
  * Peri-implant probing depth (6 points).
  * Bleeding on probing (presence or absence).
  * Suppuration on probing (presence or absence).
  * Plaque index (presence or absence).
Presence of prosthetic complications | At 6 and 12 months
  Defined as:
  * Number of maintenance visits
  * Crown screw loosening ("Yes" or "No")
  * Abutment screw loosening ("Yes" or "No")
  * Implant fracture ("Yes" or "No")
  * Crown screw fracture ("Yes" or "No")
  * Abutment screw fracture ("Yes" or "No")
  * Framework fracture ("Yes" or "No")
  * Crown ceramic chipping ("Yes" or "No")

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain